CLINICAL TRIAL: NCT04747184
Title: Variations in the Composition of Respiratory Microbiota Among Asthmatic and Non-asthmatic Subject
Brief Title: Variations in the Composition of Respiratory Microbiota
Status: Completed | Type: Observational
Sponsor: Applied Science Private University (Other)
Responsible Party: Sponsor
Other Study IDs: 1800164
Record Dates: First submitted 2021-02-04; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Asthma
Keywords: Asthma; Respiratory microbiota; Haemophilus influenzae; Oral corticosteroids; Inhalers
MeSH Terms: conditions — Asthma; Haemophilus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All participants were asked to expectorate a sputum sample in special sterile tubes indicated for sputum collection. Particular care was taken to avoid contamination of the sputum sample with the saliva and post-nasal drip by asking the participants to rinse their mouth with sterile water before inducing the sputum sample. Then the expectorated sputum specimen was immediately homogenized and stored in the deep freezer (-80°C) for DNA extraction for microbial gene sequencing and sequence analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthmatic patients: Asthmatic patients aged 14-year-old, and more were included in the study. Knowing that patient with the age of 14-year is treated as adults at Al Bashir Hospital. Smokers, patients reported to have taken antibiotics for at least two months before study enrolment, and patients who had other respiratory diseases or infections were excluded from the study.
  Interventions: Other: DNA extraction and 16S rRNA sequencing
- Healthy subjects: Healthy subjects aged 14-year-old, and more were included in the study. Smokers, patients reported to have taken antibiotics for at least two months before study enrolment, and patients who had other respiratory diseases or infections were excluded from the study.
  Interventions: Other: DNA extraction and 16S rRNA sequencing

INTERVENTIONS:
Other: DNA extraction and 16S rRNA sequencing — DNA extraction using QIAamp® DNA mini kit (QIAGEN) was done under aseptic techniques in the sterile room for all samples according to the manufacturer instructions. The DNA extracts for the 54 samples collected (27 from asthmatic patients and 27 from healthy subjects) were stored at -80° C in a sterile Eppendorf tubes until they were sent to the Molecular Research (MR DNA) Lab (Molecular Research LP, Shallowater, TX, USA) for sequencing.

SUMMARY:
Induced sputum samples were obtained from 27 asthmatic patients and 27 non-asthmatic subjects. Sequencing of the V4 region of 16S rRNA gene using Illumina MiSeq was performed, followed by analysis of alpha and beta diversity.

DETAILED DESCRIPTION:
The study was conducted over 10 months, from March to December 2019, with patients recruited from Al Bashir public hospital,A convenient sample of 54 participants were approached (27 asthmatic patients and 27 healthy subjects). All the asthmatic patients were recruited from an outpatient clinic at Al Bashir hospital. Study participants were informed about the nature of the study and were included only after obtaining their consent verbally and voluntary. Sociodemographic characteristics were collected from all study participants.

Specimens were collected according to the CDC guidelines for collecting respiratory diseases' samples. All participants were asked to expectorate a sputum sample in special sterile tubes indicated for sputum collection. Particular care was taken to avoid contamination of the sputum sample with the saliva and post-nasal drip by asking the participants to rinse their mouth with sterile water before inducing the sputum sample. Then the expectorated sputum specimen was immediately homogenized and stored in the deep freezer (-80°C) for DNA extraction for microbial gene sequencing and sequence analysis.

located in Amman, the capital city of Jordan. DNA extraction and 16S rRNA sequencing DNA extraction using QIAamp® DNA mini kit (QIAGEN) was done under aseptic techniques in the sterile room for all samples according to the manufacturer instructions. The DNA extracts for the 54 samples collected (27 from asthmatic patients and 27 from healthy subjects) were stored at -80° C in a sterile Eppendorf tubes until they were sent to the Molecular Research (MR DNA) Lab (Molecular Research LP, Shallowater, TX, USA) for sequencing. Briefly, PCR amplification of the 16s rRNA gene and its subsequent sequencing was done using Illumina. The 16s rRNA gene V4 variable region PCR primers ill27Fmod (AGRGTTTGATCMTGGCTCAG) /ill519Rmod (GTNTTACNGCGGCKGCTG) with barcode on the forward primer were used in 30 cycles using the HotStarTaq Plus Master Mix Kit (Qiagen, USA). After amplification, PCR products were checked in 2% agarose gel to determine the success of amplification and the relative intensity of bands.

The pooled and purified PCR product was then used to prepare the Illumina DNA library. Sequencing was performed on a MiSeq following the manufacturer's guidelines. Sequence data were processed using the MR DNA analysis pipeline (MR DNA, Shallowater, TX, USA). In summary, the sequences were joined, depleted of barcodes then sequences <150bp removed, sequences with ambiguous base calls were removed. Sequences were denoised, Operational taxonomic units (OTUs) generated and chimeras removed. The OTUs were defined by clustering at 3% divergence (97% similarity). Final OTUs were taxonomically classified using BLASTn against a curated database derived from RDPII and NCBI (www.ncbi.nlm.nih.gov, http://rdp.cme.msu.edu). For alpha diversity index, namely, Shannon index H, it was carried out in "Past Program" for data analysis version 4.02, after filtering out the reading with relative abundance of <1%. Shannon index varies from 0 for communities with only a single taxon to high values for communities with many taxa (DeJong, 1975).

ELIGIBILITY:
Inclusion Criteria:

1. Asthmatic patients
2. healthy subjects
3. aged 14-year-old

Exclusion Criteria:

1. Smokers
2. patients reported having taken antibiotics for at least two months before study enrolment 3- patients who had other respiratory diseases or infections.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Asthmatic, non-smoker, aged 14 years-old living in Jordan
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
To identify the common microorganisms in the LRT among asthmatic patients and non-asthmatic subjects in Jordan | 10 months
  To asses the microbiome in the LRS between asthmatic patients and non-asthmatic by sequencing the 16s rRNA gene from the collected samples, after extracting the DNA

SECONDARY OUTCOMES:
To identify a common microbial bioindicator that could be used as a diagnostic tool | 10 months
  To calculate a common microbial bioindicator that could be used as a diagnostic tool for an early diagnosis of asthma using 16s ribosomal RNA gene sequencing from sputum samples from the study population using statistical analysis and the biodiversity indicators

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Al-Najjar, PhD, Principal Investigator — Faculty of Pharmacy, Applied Science Private University
Locations (1):
- Applied Science private University, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided